CLINICAL TRIAL: NCT03749837
Title: Is a Rigid Fiberscope With a Flexible Tip Superior to Standard Flexible Fiberoptic Intubation: a Prospective Multicentre Randomised Controlled Trial
Brief Title: C-MAC Video Stylet vs. Video Endoscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018-00629
Record Dates: First submitted 2018-11-08; First posted 2018-11-21 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Intubation
MeSH Terms: interventions — Capsule Endoscopes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- C- MAC VS (Experimental): Intubation with C- MAC VS
  Interventions: Device: C- MAC VS
- Video Endoscope (Active Comparator): Intubation with standard fiberoptic scope
  Interventions: Device: Video Endoscope

INTERVENTIONS:
Device: C- MAC VS — The C-MAC VS is a new device on the airway management aid market. It will be used according to the instructions of the distributor. Before the study starts on humans, each study participants will do at least 5 intubations on an airway manikin or more until he or she feels confident to use the device.
  Arms: C- MAC VS
Device: Video Endoscope — Fiberoptic video endoscopic devices are standard aids to facilitate intubation on all study sites and are used according to the instructions to use. To facilitate fiberoptic intubation a macintosh blade to raise the root of tongue will be used. Also with these devices the study participants need at least 5 trials to intubate a manikin (or more to feel confident) before they are going to use the study device in patients.
  Arms: Video Endoscope

SUMMARY:
The purpose of the study is to compare first attempt success rates and time until intubation to establish the learning curves of the participating anaesthesiologists with two different intubation strategies: (Karl Storz C-MAC VS (Video Stylet) and the standard flexible intubation video endoscope at the study site.

DETAILED DESCRIPTION:
The intubation of the trachea is a crucial procedure in anaesthesia and emergency medicine, therefore it is considered as one of the core competences in these disciplines. Novices in the field need to learn intubation fast and without harming patients to ensure a patent airway if needed.

According to the European Union of Medical Specialists (U.E.M.S., 1050 Brussels, BE), every anaesthesiologist has to master different techniques for the airway management. One is the fiberoptic intubation in awake or asleep patients, to manage a difficult airway. For further training, these core competences need to be extended during the career, from level A (has knowledge) to level D (teaches or supervises others). As the intubation with flexible fiberoptic scopes is the gold standard for the management of a known difficult airway, the investigators want to compare this to a new technique. The use of flexible scopes do not guarantee easy intubation in every difficult airway situation and intubation sometimes is difficult to achieve and requires high proficiency (unability to steer, unability to overcome an anatomical obstacle). Various approaches were introduced by the medical device industry to overcome that problem. One new device is a rigid video stylet with a flexible tip (Karl Storz C-MAC VS), which is an advancement of the older rigid scope "Bonfils" (Karl Storz).

Intubation training with the Bonfils stylet has been shown to require about 20 consecutive tracheal intubations by novices to reach expert time. Learning curves for fiberoptic intubations seem to be similar, but a greater variance was observed. A study of the investigators research-group (unpublished data, KEK 247/09), comparing learning curves between the rigid fiberoptic Bonfils and the semi-rigid fiberoptic SensaScope suggested a 90% success rate for intubation within 60 seconds after about 15 trials (Bonfils) and 20 trials (SensaScope). In comparison, there is no validated data for the use of rigid scopes with flexible tips, as these tool are very new.

Video stylets are tools originally designed for difficult airway management as well. The C-MAC VS combines rigid and semi-rigid abilities. Intubation seems to become very easy. But yet, there is no data available which proves that assumption. Thus the study wants to evaluate if intubation success and time is superior with the C-MAC Video Scope compared to the difficult intubation gold standard, the intubation with a standard flexible fiberoptic scope.

ELIGIBILITY:
Inclusion Criteria:

* Anaesthesiologists starting in the respective anaesthesia department who are not experienced with tracheal intubation with the study devices
* Informed Consent as documented by signature (Appendix Informed Consent Form)
* Novice to the C-MAC VS
* No/few fiberoptic oral asleep intubation experience (max. 5x during the last year)

Exclusion Criteria:

* More than 5 uses during the past year of either one of the study devices
* Not available at the study site during entire study (expected drop outs)
* Not able to fill out English case reports
* Patients: Planned delayed extubation (e.g. planned transfer to ICU)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Time (seconds) to successful orotracheal intubation during the first successful attempt. | Start: Device passes patients lips; End: Device is completely removed out of the tracheal tube (a trial consists of a maximum of 2 intubation attempts, each with a maximum duration of 120 seconds)
  With the C-MAC VS and the standard flexible scope

SECONDARY OUTCOMES:
Overall time from startpoint to glottic view | It cannot be longer than 240 seconds and is defined for unsuccessful trials, i.e. if no intubation was established, as 360 seconds.
  The overall time is defined as the total time to glottic view, summarized over all attempts.
Time to first end expiratory CO2 reading | Start: Device passes patients lips; End: First end expiratory CO2 reading (trial in total not >240 seconds)
  After the airway is secured the first end expiratory CO2 is shown.The investigators will use the standard non-invasive monitoring of the University Hospital to measure the end expiratory CO2
Number of intubation attempts | Start: Device passes patients lips; End: Device is completely removed out of the tracheal tube (trial in total not >240 seconds)
  End of an attempt defined as: device has to be completely removed out of the patient's airway.
Subjective difficulty of the intubation procedure | Start: Device passes patients lips; End: Device is completely removed out of the tracheal tube (trial in total not >240 seconds
  The VAS- Visual analogue scale (score 1-10) is used. It is a measurement instrument for subjective characteristics that cannot be directly measured. Therefore numbers are used to evaluate.
Cormack/Lehane grade | Start: Device passes patients lips; End: Device is completely removed out of the tracheal tube (trial in total not >240 seconds)
  The Cormack/Lehane grade is used to describe the laryngeal view during laryngoscopy. It is rated by the supervisor.
Limited or restricted vision through the devices (either C MAC VS or a standard flexible scope) | Start: Device passes patients lips; End: Device is completely removed out of the tracheal tube (trial in total not >240 seconds)
  The view can be clear or blurred.
Correlation to patients' anatomical characteristics | Start: Device passes patients lips; End: Device is completely removed out of the tracheal tube (trial in total not >240 seconds)
  To assess the influence of difficulty with the airway
Patients vital parameter such as heart rate, during the intubation attempt | Start: Device passes patients lips; End: Device is completely removed out of the tracheal tube (trial in total not >240 seconds)
  The investigators will use the standard non-invasive monitoring of the University Hospital to measure the heart rate.
Patients vital parameter such as blood pressure, during the intubation attempt | Start: Device passes patients lips; End: Device is completely removed out of the tracheal tube (trial in total not >240 seconds)
  The investigators will use the standard non-invasive monitoring of the University Hospital to measure the blood pressure (in millimeters of mercury)
Patients vital parameter such as oxygen saturation, during the intubation attempt | Start: Device passes patients lips; End: Device is completely removed out of the tracheal tube (trial in total not >240 seconds)
  The investigators will use the standard non-invasive monitoring of the University Hospital to measure the oxygen saturation (SpO2 in percent).
Participants characteristics and demographic data | Before the study session starts (up to 24 hours before the first intubation attempt)
  Basic demographic data (including years of experience in anaesthesia).
Patients demographic data such as height | During the process of screening, up to 24 hours before the study session starts
  The size of each patient will be presented in meter/centimeter
Patients demographic data such as weight | During the process of screening, up to 24 hours before the study session starts
  The weight of each patient will be presented in kilograms
Patients demographic data such as ASA risc classification (ASA= American Society of Anaesthesiologists) | During the process of screening, up to 24 hours before the study session starts
  The ASA grading system is used to evaluate the degree of a patient's physical state before selecting the anesthetic or before performing surgery.
Patients demographic data such as age | During the process of screening, up to 24 hours before the study session starts
  The age of each patient will be presented in years.
Patients demographic data such as gender | During the process of screening, up to 24 hours before the study session starts
  The gender of each patient will be presented in female or male.

OTHER OUTCOMES:
Incidence of injuries due to intubation attempts | Follow-Up on the first post anaesthesia day (maximum 24 hours post anaesthesia)
  Dental damage, mucosal damage, hoarseness, sore throat, swallowing disorders
How often a "hand over to specialist" happens | Start: Device passes patients lips; End: Device is completely removed out of the tracheal tube (trial in total not >240 seconds)
  The device has to be handed over to the supervisor

CONTACTS AND LOCATIONS:
Overall Officials: Lorenz Theiler, Prof., M.D, Principal Investigator — Department of Anaesthesiology and Pain Therapy
Locations (3):
- LHSC / St. Joesephs, London, Ontario, Canada
- Miguel Servet University Hospital, Zaragoza, Spain
- Inselspital, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kleine-Brueggeney M, Greif R, Urwyler N, Wirthmuller B, Theiler L. The performance of rigid scopes for tracheal intubation: a randomised, controlled trial in patients with a simulated difficult airway. Anaesthesia. 2016 Dec;71(12):1456-1463. doi: 10.1111/anae.13626. Epub 2016 Sep 27. PMID 27670928
- [Background] Halligan M, Charters P. A clinical evaluation of the Bonfils Intubation Fibrescope. Anaesthesia. 2003 Nov;58(11):1087-91. doi: 10.1046/j.1365-2044.2003.03407.x. PMID 14616594
- [Background] Isono S, Greif R, Mort TC. Airway research: the current status and future directions. Anaesthesia. 2011 Dec;66 Suppl 2:3-10. doi: 10.1111/j.1365-2044.2011.06928.x. PMID 22074073
- [Background] Levitan RM, Goldman TS, Bryan DA, Shofer F, Herlich A. Training with video imaging improves the initial intubation success rates of paramedic trainees in an operating room setting. Ann Emerg Med. 2001 Jan;37(1):46-50. doi: 10.1067/mem.2001.111516. PMID 11145770
- [Background] Sakles JC, Chiu S, Mosier J, Walker C, Stolz U. The importance of first pass success when performing orotracheal intubation in the emergency department. Acad Emerg Med. 2013 Jan;20(1):71-8. doi: 10.1111/acem.12055. PMID 23574475
- [Background] Dalal PG, Dalal GB, Pott L, Bezinover D, Prozesky J, Bosseau Murray W. Learning curves of novice anesthesiology residents performing simulated fibreoptic upper airway endoscopy. Can J Anaesth. 2011 Sep;58(9):802-9. doi: 10.1007/s12630-011-9542-2. Epub 2011 Jun 28. PMID 21710368
- [Background] Smith JE, Jackson AP, Hurdley J, Clifton PJ. Learning curves for fibreoptic nasotracheal intubation when using the endoscopic video camera. Anaesthesia. 1997 Feb;52(2):101-6. doi: 10.1111/j.1365-2044.1997.23-az023.x. PMID 9059089